CLINICAL TRIAL: NCT03286452
Title: Real-World Effectiveness Study of PuraPly™ AM on Wounds
Brief Title: The RESPOND Registry
Acronym: RESPOND
Status: Completed | Type: Observational
Sponsor: Organogenesis (Industry)
Collaborators: Continuum Clinical Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 16-REG-002-PPAM
Record Dates: First submitted 2017-08-26; First posted 2017-09-18 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Partial Thickness Wound; Pressure Ulcer; Venous Ulcer; Diabetic Ulcer; Surgical Wounds; Trauma Wounds; Draining Wounds; Chronic Vascular Ulcer
Keywords: Antimicrobial; Collagen; Bioburden; Biofilm; PHMB; Chronic wounds; Acute wounds
MeSH Terms: conditions — Pressure Ulcer; Varicose Ulcer; Surgical Wound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: PuraPly™ Antimicrobial Wound Matrix — PuraPly™ Antimicrobial Wound Matrix consists of a collagen sheet coated with 0.1% polyhexamethylenebiguanide hydrochloride (PHMB) intended for the management of wounds.
  Other Names: PuraPly™ Antimicrobial; PuraPly™ AM

SUMMARY:
The RESPOND Registry is an observational study to assess the impact of PuraPly™ AM on the management of wounds in real world clinical settings; no experimental intervention is involved.

DETAILED DESCRIPTION:
The purpose of this study is to assess the impact of PuraPly™ AM on the management of wounds in real world clinical settings as it leads to an improvement in wound bed condition (i.e increase in healthy granulation tissue, reduction in bioburden, and reduction in amount of exudate).

The RESPOND Registry is a prospective, non-interventional research initiative to collect information on patients who are eligible to receive PuraPly™ AM, and no interventional procedures will be mandated by this protocol.

Enrolled and eligible patients will receive standard wound care clinical assessments and any additional care as determined by the treating wound care clinician. Although multiple wounds may be treated simultaneously, one wound will be identified as the target wound, and characteristics regarding this wound will be consistently documented.

The case series is being undertaken to better understand PuraPly™ AM utilization and subsequent healing outcomes as well as to evaluate the effects of concomitant wound therapy on healing. Patient's participation may involve follow-up for up to 24 weeks following application of PuraPly™ AM.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient, or their legally authorized representative (LAR), has read, understood and signed and Institutional Review Board (IRB) approved Informed Consent Form (ICF).
* Patient has a wound appropriate for receiving PuraPly™ AM, including:

  * Partial or full-thickness wound
  * Pressure ulcer
  * Venous ulcer
  * Diabetic ulcer
  * Chronic vascular ulcer
  * Tunneled/undermined wound
  * Surgical wound (e.g., donor sites/graft, post-Mohs' surgery, post-laser surgery, podiatric surgery wound, wound dehiscence)
  * Trauma wound (abrasions, lacerations, second degree burns, and skin tears)
  * Draining wound

Exclusion Criteria:

* Patient has a known sensitivity to porcine materials.
* Patient has a third-degree burn.
* Patient has a known sensitivity to polyhexamethylenebiguanide hydrochloride (PHMB).
* Patient's target wound was previously treated with PuraPly™ AM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 300 patients to be enrolled by approximately 30 US-based Physician Investigators. Patients are male or female at least 18 years old, with an eligible target wound that meets the Investigator's wound specific treatment goals; including the management of bioburden, support of granulation tissue formation, and support of wound closure.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2019-01-26 (Actual)

PRIMARY OUTCOMES:
Reduction in size of wound area | Up to 24 weeks
  As measured from change in size from baseline
Time to complete wound closure | Up to 24 weeks
  As measured by time to complete wound closure from baseline
Improvement in wound bed condition | Up to 24 weeks
  As measured from change in status from baseline

SECONDARY OUTCOMES:
Improvement in patient reported pain | Up to 24 weeks
  As measured change in status from baseline as assessed by the PAIN visual analogue scale (PAIN-VAS)
Improvement in patient reported quality of life | Up to 24 weeks
  As measured by change in status from baseline as assessed by the SF-12 QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Teichman, DPM, Principal Investigator — PA Foot and Ankle Association; Shaun Carpenter, M.D., Principal Investigator — Wound Care Associates, LLC.; Daniel L Kapp, M.D., Principal Investigator — Jupiter Medical Center; Kerry Thibodeaux, M.D., Principal Investigator — Opelousas General Hospital Wound Center; George Koullias, M.D., Principal Investigator — Southampton Hospital; Raymond Abdo, DPM, Principal Investigator — Saint Louis Foot and Ankle; Barry Wisler, DPM, Principal Investigator — Robert Wood Johnson Hamilton; Carlos Trabanco, MD, Principal Investigator — West Gables Rehabilitation Hospital; Ifat Kamin, MD, Principal Investigator — Meriter Hospital Inc., DBA: UnityPoint Health Heart and Vascular Institute; Amanda Estapa, NP, Principal Investigator — Institute for Advanced Wound Healing; Northshore Specialty Hospital; Michael Menack, MD, Principal Investigator — CentraState Medical Center; Ritu Gothwal, MD, Principal Investigator — Advanced Wound Care Center at Yavapai Regional Medical Center; Mark Iafrati, MD, Principal Investigator — Tufts Medical Center; Paula Pons, MD, Principal Investigator — Saint Joseph's Center for Wound Care and Hyperbaric Medicine; Taysha Howell, MD, Principal Investigator — Oklahoma Wound Center; Allan Grossman, DPM, Principal Investigator — Harrisburg Foot and Ankle Center, Inc.
Locations (15):
- United States (15):
  - Advanced Wound Care Center at Yavapai Regional Medical Center, Prescott Valley, Arizona
  - Jupiter Medical Center, Jupiter, Florida
  - West Gables Rehab Hospital, Miami, Florida
  - Institute for Advanced Wound Healing; Northshore Specialty Hospital, Covington, Louisiana
  - Wound Care Associates, LLC., Hammond, Louisiana
  - Opelousas General Hospital Wound Center, Opelousas, Louisiana
  - Saint Louis Foot and Ankle, St Louis, Missouri
  - CentraState Medical Center, Freehold, New Jersey
  - Robert Wood Johnson Hamilton, Hamilton, New Jersey
  - Southampton Hospital, Southampton, New York
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Sacred Heart Hospital, Allentown, Pennsylvania
  - Harrisburg Foot and Ankle Center, Inc., Harrisburg, Pennsylvania
  - Greensville Health System, Greenville, South Carolina
  - Meriter Hospital Inc., DBA: UnityPoint Health Heart and Vascular Institute, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bain MA, Koullias GJ, Morse K, Wendling S, Sabolinski ML. Type I collagen matrix plus polyhexamethylene biguanide antimicrobial for the treatment of cutaneous wounds. J Comp Eff Res. 2020 Jul;9(10):691-703. doi: 10.2217/cer-2020-0058. Epub 2020 Jun 1. PMID 32476449